CLINICAL TRIAL: NCT06832800
Title: Modified Diagnosis and Treatment of Neonatal Hemolysis Incorporated With ETCOc Measurement in Severe Neonatal Hyperbilirubinemia Management
Brief Title: Modified Diagnosis and Treatment of Neonatal Hemolysis With ETCOc in sNH
Acronym: MDTinsNH
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO2024-737; 2025KY929 (Other: The Medical and Health Research Project of Zhejiang Province)
Record Dates: First submitted 2025-01-31; First posted 2025-02-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: ETCOc; neonatal hemolysis; neonatal hyperbilirubinemia; modified
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Experimental): modified diagnosis and treatment (MDT) for neonatal hemolysis
  Interventions: Combination Product: MDT
- control (Other): Control (current) method for sNH (severe neonatal hemolysis) with the description as follow：
  1. Diagnosis of neonatal hemolysis： The neonatal subjects with symptom of hyperbilirubinemia are diagnosed as hemolysis if they have positive Direct Antiglobulin Test (DAT) or positive release test result.
  2. Exchange transfusion (ET) therapy for sNH： The neonatal subjects with symptom of hyperbilirubinemia are treated with ET therapy if their Total serum bilirubin (TSB) reaches or exceeds the current exchange transfusion threshold;
  Interventions: Other: control (current management)

INTERVENTIONS:
Combination Product: MDT — （actually not combination product, but have to select that option in order to delete warning in "study desine"）MDT method for sNH with the description as follow： 1. diagnosis of neonatal hemolysis：
  The neonatal subjects with symptom of hyperbilirubinemia are diagnosed as hemolysis if they met one criterion from Category A or two criteria from Category B:
  Category A:
  1. Positive DAT
  2. Significantly elevated ETCOc;
  3. Significant morphological abnormalities
  Category B:
  1. Positive release test;
  2. Elevated ETCOc;
  3. COHb > 1.2%;
  4. Hb < 140 g/L or Hct) < 40%;
  5. Ret > 6%. 2.Exchange transfusion (ET) therapy for sNH： any of the following criteria are met:
  (1) TSB ≥ the current ET threshold; (2) TSB > (ET - 2) mg/dL or the increase of TSB > 0.5 mg/dL/h, accompanied by abnormal aEEG findings; (3) TSB > (ET - 2) mg/dL or > 0.5 mg/dL/h, accompanied by a BIND score of 4-6; (4) Presence of clinical manifestations of acute ABE; (5) BIND score of 7-9.
  Arms: study
Other: control (current management) — Control (current) method for sNH (severe neonatal hemolysis) with the description as follow：
  1. Diagnosis of neonatal hemolysis： The neonatal subjects with symptom of hyperbilirubinemia are diagnosed as hemolysis if they have positive Direct Antiglobulin Test (DAT) or positive release test result.
  2. Exchange transfusion (ET) therapy for sNH： The neonatal subjects with symptom of hyperbilirubinemia are treated with ET therapy if their Total serum bilirubin (TSB) reaches or exceeds the current exchange transfusion threshold;
  Arms: control

SUMMARY:
The goal of this clinical trial is to learn if modified diagnosis and treatment (MDT) of neonatal hemolysis (a common cause to newborn jaundice) incorporated with ETCOc measurement (a non-invasive measurement of exhaled gas) works to prevent brain damage in newborns with severe hyperbilirubinemia (sNH). It will also learn about the. occurrence of cranial MRI in the study participants. The main questions it aims to answer are:

* Does MDT lower the possibilities participants have brain damage before the age of one?
* How many times of abnormalities in cranial MRI is detected before the age of one? Researchers will compare MDT to a control (a current management) to see if MDT works to prevent brain damage in newborns with sHN.

Participants will:

* Take MDT or a control method in the management of sNH
* Assess if there's brain damage before discharge and at the year of one
* Record how many times of abnormalities in cranial MRI is detected before the age of one

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria:

Infants with gestational age of 35(+0) to 41(+6) weeks and birth weight ≥ 2500 grams

* Infants with severe neonatal hyperbilirubinemia, including those whose serum total
* bilirubin (TSB) levels reach above 20 mg/dL or whose TSB levels at any time reach within 2 mg/dL of the exchange transfusion threshold (i.e., TSB > (threshold - 2) mg/dL).

Exclusion Criteria:

* Infants with definite congenital genetic metabolic diseases, chromosomal or genetic disorders, or severe malformations.

Ages: 4 Hours to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
neural damage confirmed by professional assessments such as Bayley Scales | at the age of 12 months
  Neurological impairment, including any of the following: diagnosis of cerebral palsy, diagnostic hearing tests indicating hearing impairment, or a score lower than 85 on the Bayley Scales Neurobehavioral Assessment. Bayley Scales means Bayley Scales of Infant and Toddler Development and it can assess the neural development of infants including Cognitive, Language (Receptive/Expressive), Motor (Fine/Gross), Social-Emotional, and Adaptive Behavior. Standard scores for each domain range from 40 to 160 (mean = 100; SD = 15). Higher scores indicate better developmental outcomes, while lower scores suggest potential delays.
  For example, a cognitive score of 115 reflects performance above the average range, whereas a score of 85 falls below the average range.

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Bao, Doctor, Principal Investigator — Women's Hospital, Zhejiang University School of Medicine; Bao, Doctor, Principal Investigator — Women's Hospital, Zhejiang University School of Medicine
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Yes